CLINICAL TRIAL: NCT00001850
Title: Evaluation of Women and Men With Endocrine and Reproductive-Related Conditions
Brief Title: Evaluation of Women With Endocrine and Reproductive-Related Conditions
Status: Terminated | Type: Observational
Why Stopped: Terminated at the direction of the NIH IRBO.
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990103; 99-CH-0103
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Endocrine Disease; Infertility; Leiomyoma; Endometriosis; Fibroids
Keywords: Reproductive Surgery; Infertility; Hormone Replacement Therapy; GATA 2; Sickle Cell; Natural History
MeSH Terms: conditions — Endocrine System Diseases; Infertility; Leiomyoma; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children: with reproductive disorders
- Men: with reproductive disorders
- Woman: with reproductive disorders

SUMMARY:
This study was designed to allow inpatient and outpatient evaluation of women with a variety of reproductive and endocrine-related disorders for purposes of research and physician education.

The evaluations may include ultrasound examinations, blood, saliva, and/or urine samples. In some cases, specific laboratory or X-ray studies will be performed to confirm the diagnosis or assist in the treatment of the patient. These additional tests will be conducted within the guidelines of current gynecologic practice. In some cases, the patient will receive medical or surgical treatment for their disorder.

The purpose of this study is to provide an opportunity for physicians to evaluate women with medical conditions of reproduction. These evaluations and treatments will support clinical training and research for the accredited training program in reproductive endocrinology at the National Institute of Child Health and Human Development (NICHD).<TAB>

DETAILED DESCRIPTION:
The specific objective of this protocol is to gain knowledge and collect data in order to allow for hypothesis generation in future research as well as give NICHD investigators and trainees hands on experience related to the diagnoses, management, treatment and follow-up of reproductive endocrine disorders. Such disorders include but are not limited to Polycystic ovarian syndrome, Endometriosis, Primary ovarian insufficiency, Recurrent pregnancy loss, Primary amenorrhea and Infertility. This information will be taken from standard medical care/procedures and follow up of patients and healthy volunteers. It allows investigation into the problems of these patients for the purpose of furthering general knowledge and teaching.

ELIGIBILITY:
* Inclusion Criteria:
* Subjects aged 1-85 with reproductive endocrine related conditions.
* Young women, women of reproductive age, and older women are the focus of this protocol.
* Girls with reproductive disorders under the age of 18 will be studied and their assent will be obtained if possible along with the consent of their parent/guardian.
* Reproductive disorders of men will be included.

Exclusion Criteria:

* Pregnant women over 23 weeks will be excluded, since there are no on-campus prenatal or neonatal facilities. If we see patients in consultation after 23 weeks, as is our practice, we will provide a report to the referring PI on that protocol as well as the patient's personal obstetrician. We do not provide long term obstetrical care.
* Patients specifically requesting in vitro fertilization will not be considered candidates and will not be seen under this protocol. These patients may be seen for a consultation, but will be referred for these services outside of the NIH.
* Pregnant patients requiring fetal surgery will be excluded since there are no on-campus neonatal facilities.

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 1-85 with reproductive disorders
Sampling Method: Non-Probability Sample
Enrollment: 833 (Actual)
Dates: Start 1999-05-10 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
To provide a mechanism for reproductive endocrine fellows and staff to evaluate woman with medical conditions of interest for fellow training and clinical training and education. | 11/30/2025
  To provide a mechanism for reproductive endocrine fellows and staff to evaluate woman with medical conditions of interest for fellow training and clinical training and education.

CONTACTS AND LOCATIONS:
Overall Officials: Alan H DeCherney, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-CH-0103.html